CLINICAL TRIAL: NCT05339412
Title: Technology-based Training Tool for an Empirically-Supported Group-Based HIV and STI Prevention Intervention for Juvenile Offenders
Brief Title: Technology-based Training Tool for PHAT Life
Acronym: PhatLife-II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Research Behavioral Intervention Strategies, Inc. (Industry)
Collaborators: University of Illinois at Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MD014113-02
Record Dates: First submitted 2022-02-28; First posted 2022-04-21 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: HIV Infection; Sexually Transmitted Infections; Implementation
MeSH Terms: conditions — HIV Infections; Sexually Transmitted Diseases

STUDY DESIGN:
Intervention Model Description: Participants are randomized to one of two conditions: (1) technology based training tool only; or (2) technology based training tool plus live supervision.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Technology Based Training Tool Only (Experimental): The technology-based training tool will train facilitators to deliver the behavioral health intervention PHAT Life, which is an innovative HIV/STI, substance use, and mental health intervention for juvenile offenders. The training tool reviews each of PHAT Life's 8 sessions. The curriculum targets broad psychosocial factors implicated in HIV/STI-risk behavior, including promoting positive attitudes toward HIV/STI prevention, self-efficacy to reduce risk, and less substance misuse and sexual risk taking. Content emphasizes the importance of emotion regulation skills to manage strong feelings, uses goal setting and training in positive thought processes to plan ahead, encourages recognition of personal responsibility in future outcomes, and helps youth identify strategies and behaviors to accomplish short- and long-term goals.
  Interventions: Behavioral: Training Tool for Preventing HIV/AIDS among Teens (PHAT) Life
- Technology Based Training Tool plus Live Supervision (Experimental): Participants randomized to this condition will receive (in addition to the training tool described above) access to live supervision delivered remotely via commercially available video conferencing software (Zoom). Facilitators-in-training will complete two mock roleplays of curriculum activities, which can be conducted live via Zoom with PHAT Life trainers (either Dr. Floyd or Dr. Snow-Hill) or can be recorded and submitted via the app. Trainers will review for fidelity and provide feedback. During the supervision sessions, participants will have the opportunity to clarify content, ask questions, roleplay group sessions to practice difficult parts of the group sessions, and review feedback on role plays.
  Interventions: Behavioral: Training Tool for Preventing HIV/AIDS among Teens (PHAT) Life

INTERVENTIONS:
Behavioral: Training Tool for Preventing HIV/AIDS among Teens (PHAT) Life — The technology-based training tool will train facilitators to deliver the behavioral health intervention PHAT Life, which is an innovative HIV/STI, substance use, and mental health intervention for juvenile offenders. The training tool reviews each of PHAT Life's 8 sessions. The curriculum targets broad psychosocial factors implicated in HIV/STI-risk behavior, including promoting positive attitudes toward HIV/STI prevention, self-efficacy to reduce risk, and less substance misuse and sexual risk taking. Content emphasizes the importance of emotion regulation skills to manage strong feelings, uses goal setting and training in positive thought processes to plan ahead, encourages recognition of personal responsibility in future outcomes, and helps youth identify strategies and behaviors to accomplish short- and long-term goals.

SUMMARY:
Youth under age 18 involved in the criminal justice system are disproportionately minorities & affected by substance abuse, mental illness, & HIV/STI. Most young offenders are released on community supervision without the STI, mental health, or substance use screening, diagnosis, & treatment afforded detained youth, despite similar rates of risk behavior. Their long-term trajectory is poor, costs to society are high, & lasting effects on community well-being & individual employment prospects are profound. Altering this trajectory is a public health priority. Preventing HIV Among Teens (PHAT) Life is an evidence-based program that meets the need in juvenile justice to address youths' co-morbid health problems. The next step in ensuring that this decade-long line of research produces actual, real-world improvements in the lives of probation youth is to develop a PHAT Life training strategy that is effective, cost-effective, & sustainable within juvenile justice settings. The private/public collaboration between ORBIS & UIC will leverage existing resources & competencies to create a commercially viable technology-based training tool for PHAT Life with great potential for sustainability & cost-effectiveness. This Phase II uses a formative process to refine, enhance & complete the technology-based training tool to include: (a) an interactive multimedia web browser & mobile application, (b) dynamic multimedia presentations & interactive queries, (c) video examples of mock intervention delivery, (d) audio narration along with scripted language, (e) brief quizzes to ensure comprehension & knowledge acquisition, (f) opportunities to "learn more" by clicking on tabs for supplemental information, (g) targeted referrals to appendix materials, (h) games to promote engagement, & (i) other adaptations based on Phase I feedback. The proposed technology-based training tool should be highly sustainable, because it (a) relies on "indigenous" personnel to deliver the intervention, (b) is likely to prove cost-effective since it will utilize a technology that can deliver training at scale, & (c) will improve fidelity by leveraging technology to provide consistent training experiences to para-professionals. The training tool will be evaluated via a 2-arm RCT with 130 individuals who work with justice-involved youth. Trainees will receive the technology-based training tool.

DETAILED DESCRIPTION:
This study will comply with the NIH Policy on the Use of sIRB for Multi-Site Research. The University of Illinois Chicago (UIC) has been selected to serve as the single IRB of record (sIRB) for the research described in this proposal. Once the PHAT Life Training Tool is complete, Investigators will enroll 6 paraprofessionals to conduct a brief usability test to ensure the tool is working properly. After edits are made based on the feedback from the usability test, 10 paraprofessionals who work with justice-involved youth will pilot test the study materials and protocol to ensure that Investigators are ready for scale in a randomized trial. To meet the proposed study's aims, the research team has commitment from three sites who serve justice-involved youth (see Letters of Support): (a) Cook County Juvenile Temporary Detention Center, (b) Cook County Department of Probation and Court Services, and (c) Heartland Alliance. Together, there are about 445 eligible staff across settings. The proposed sample (N=130) represents 29% of eligible participants. Investigators, thus, expect minimal difficulty reaching the proposed sample size. Researchers will present the project at agency staff meetings and invite people to indicate interest. Flyers will be posted in relevant spaces with researcher contact information. Researchers will offer to present information about the project at agency events. Agency staff will distribute recruitment materials to eligible personnel (e.g., probation staff or public health educators) and invite them to contact the researchers. The agency staff will also invite individuals to consent to release their contact information for the research team to contact them directly. The recruitment coordinator will contact interested individuals by phone, email, text, and instant messenger. Recruitment will continue in this manner until enrollment goals are met for each condition.

Once enrolled in the study, participants will be assigned a unique, de-identifiable project ID number, which will be affiliated with their baseline survey, Training Tool, and post-training survey. Research staff will fully explain the study and ask for their consent to participate. Participants will indicate their consent via project webpage just prior to the baseline assessment. Participants will be randomized to condition after completing their baseline measures via Qualtrics. A table will be created based on a computer-generated random numbers list that will be used by research staff to assign condition. Participants will then be provided with their login information and instructions for accessing the PHAT Life Training Tool. For those in the Training Tool Plus Supervision condition, participants will receive individualized supervision and participate in two mock role-plays of PHAT Life activities after completing the training tool. All participants will be sent the post-training assessments via Qualtrics. Finally, participants will be instructed to lead one PHAT Life group where they will audio record sessions 1 and 4 of the PHAT Life curriculum.

ELIGIBILITY:
Inclusion Criteria:

* Any staff at the recruitment sites who provides services to justice-involved youth will be eligible for this study
* Given that the training and curriculum are only offered in English, English-speaking will be an inclusion criterion

Exclusion Criteria:

• Unable to speak English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2024-01-26 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Change over time in HIV knowledge needed for HIV prevention | Baseline
  The Human Immunodeficiency Virus Knowledge Questionnaire (HIV-KQ) is an 12-item true/false measure developed to assess knowledge needed for HIV prevention. Total scores are calculated by the number of correct items. The minimum score is "0" and the maximum score is "12". A higher score indicate higher HIV knowledge.
Change over time in HIV knowledge needed for HIV prevention | Post-training (6-weeks)
  The Human Immunodeficiency Virus Knowledge Questionnaire (HIV-KQ) is an 12-item true/false measure developed to assess knowledge needed for HIV prevention. Total scores are calculated by the number of correct items. The minimum score is "0" and the maximum score is "12". A higher score indicate higher HIV knowledge.
Change over time in STI knowledge needed for HIV prevention | Baseline
  The HIV Sexually Transmitted Infections Knowledge Questionnaire (HIV-STI-KQ) is an 12-item true/false measure developed to assess knowledge needed for HIV prevention. Total scores are calculated by the number of correct items. The minimum score is "0" and the maximum score is "12". A higher score indicate higher STI knowledge.
Change over time in STI knowledge needed for HIV prevention | Post-training (6-weeks)
  The HIV Sexually Transmitted Infections Knowledge Questionnaire (HIV-STI-KQ) is an 12-item true/false measure developed to assess knowledge needed for HIV prevention. Total scores are calculated by the number of correct items. The minimum score is "0" and the maximum score is "12". A higher score indicate higher STI knowledge.
Fidelity | Post-training (6-weeks)
  The Investigators will assess treatment fidelity with self-report and audio recordings of adherence and competence. Adherence measures will determine whether the program was delivered as planned, and competence ratings will indicate the quality of intervention delivery. After each session, participants will rate whether they delivered each activity (yes/no). On a Likert scale, they will indicate how smoothly the session went, how well they knew and delivered the material, their comfort with participants, and how well the participants interacted. Open-ended questions will offer opportunities to report challenges or barriers encountered during the session. The observers will rate whether each task was completed (yes/no), and using a Likert scale (0=not very well to 5=excellent): (1) facilitator leadership skills (e.g., explained each activity correctly, was open and non-judgmental); and (2) facilitator adherence and competence on delivery of session-specific activities.

SECONDARY OUTCOMES:
Sex Education Confidence Scale | Baseline
  The Sex Education Confidence Scale (SECS) is a 22-item measure and was designed to assess how comfortable one is teaching sex education on a 6-point Likert scale. Total scores include averaging across responses. The minimum score is "1" and the maximum score is "6". A higher score indicates more confidence providing sex education.
Sex Education Confidence Scale | Post-training (6-weeks)
  The SECS is a 22-item measure and was designed to assess how comfortable one is teaching sex education on a 6-point Likert scale. Total scores include averaging across responses. The minimum score is "1" and the maximum score is "6". A higher score indicates more confidence providing sex education.
Satisfaction with Technology-Based Training | Post-training (6-weeks)
  An adapted version of the satisfaction measure currently used for the PHAT Life in-person trainings will be used to measure satisfaction with the technology-based training. This is a 21-item measure on a 5-point Likert scale. Scores are averaged across items.
Implementation Outcomes | Post-training (6-weeks)
  The implementation outcomes has 5 series of measures adapted based on the RE-AIM framework. All scores are averaged across subscales.
  1. Adoption, 12-item measure on 5-point Likert scale. Minimum (Min) score is 1 and maximum (Max) score is 5. A higher score indicates greater support for adopting the intervention;
  2. Implementation, 5-item measure on 10-point scale. Min score is 1 and Max score is 10. A higher score indicates greater support for implementing the intervention;
  3. Acceptability, 6-item measure on 4-point scale. Min score is 1 and Max score is 4. A higher score indicates greater acceptability of the intervention;
  4. Appropriateness, 5-item measure on 4-point Likert scale. Min score is 1 and Max score is 4. A higher score indicates greater beliefs that the intervention is appropriate; And
  5. Maintenance, 6-item measure on 7-point scale. Min score is 1 and Max score is 7. A higher score indicates greater support for maintaining the intervention.
Utilization: Number of Sessions | Post-training (6-weeks)
  The number of sessions logged into the website or app for each user will be evaluated using standard back-end usage data recorded by computer program.
Utilization: Total Time On-line | Post-training (6-weeks)
  The total time spent on the website or app for each user will be evaluated using standard back-end usage data recorded by computer program.
Utilization: Number of Homework Modules Completed | Post-training (6-weeks)
  The number of homework modules completed on the website or app for each user will be evaluated using standard back-end usage data recorded by computer program.
Utilization: Number of External Resources Accessed | Post-training (6-weeks)
  The number of external resources accessed for each user through the website or app will be evaluated using standard back-end usage data recorded by computer program.
Utilization: Time of Day at Log On | Post-training (6-weeks)
  The time of day initial log on to the website or app for each user will be evaluated using standard back-end usage data recorded by computer program.
Utilization: Number of Times Logged on Each Week | Post-training (6-weeks)
  The number of time logged on to the website or app each week for each user will be evaluated using standard back-end usage data recorded by computer program.
Utilization: Length of time spent in (a) information; (b) support; (c) video; (d) assessment areas of training website | Post-training (6-weeks)
  The length of time spent in each of the following training areas of the website, (a) information; (b) support; (c) video; (d) assessment, for each user will be evaluated using standard back-end usage data recorded by computer program.
Training Tool Cost Data | Post-training (6-weeks)
  Cost data will examine the relative costs of the PHAT Life training tool delivered with supervision vs. without supervision. Total cost will be calculated for (a) training tool alone and (b) training tool plus supervision versions (ΣCi for each version) divided by the average participant cost (ΣCi/n).

CONTACTS AND LOCATIONS:
Overall Officials: David R Smith, PhD, Principal Investigator — Oregon Research Behavioral Intervention Strategies, Inc.
Locations (1):
- Oregon Research Behavioral Intervention Strategies, Inc., Springfield, Oregon, United States